CLINICAL TRIAL: NCT04574713
Title: Candesartan for Migraine Prevention: A Multicentre, Binational, Triple Blind, Placebo Controlled, Parallel Group Study of Two Doses of Candesartan (8 and 16 mg)
Brief Title: Candesartan for Migraine Prevention:
Acronym: CandMig-3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Nordlandssykehuset HF (Other); Molde Hospital (Other); Haukeland University Hospital (Other); Sorlandet Hospital HF (Other Government); University Hospital, Akershus (Other); Ullevaal University Hospital (Other); Rikshospitalet University Hospital (Other); University Hospital of North Norway (Other); Tartu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 63527; 2019-003386-18 (EudraCT Number); NFR 288699. (Other Grant/Funding Number: Research Council of Norway)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Migraine
Keywords: Prevention and Control; Candesartan
MeSH Terms: conditions — Migraine Disorders | interventions — candesartan

STUDY DESIGN:
Intervention Model Description: A multicentre, binational, triple blind, placebo controlled, parallel group study of two doses
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Candesartan 8 mg (Experimental)
  Interventions: Drug: Candesartan Oral Tablet 8 mg
- Candesartan 16 mg (Experimental)
  Interventions: Drug: Candesartan Oral Tablet 16 mg
- Control group (Placebo Comparator)
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Candesartan Oral Tablet 8 mg — 1 over-encapsulated tablet once daily, containing candesartan 8 mg, for 12 weeks (84 days).
  Arms: Candesartan 8 mg
Drug: Candesartan Oral Tablet 16 mg — 1 over-encapsulated tablet once daily, containing candesartan 16 mg, for 12 weeks (84 days).
  Arms: Candesartan 16 mg
Drug: Placebo oral tablet — 1 over-encapsulated tablet once daily, containing placebo, for 12 weeks (84 days).
  Arms: Control group

SUMMARY:
The main objective of this study is to see whether the favorable preventative effect of candesartan 16 mg per day in episodic migraine, that was found previously in two smaller randomized controlled cross-over studies, can be confirmed in a larger, multicenter, randomized controlled parallel group study. In addition it will be investigated whether 1) also a smaller dose of 8 mg is effective, and 2) whether the favorable side effect profile, seen in previous studies, can be confirmed, and whether it is even better with the smaller dose.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Episodic migraine with or without aura according to ICHD-3 criteria
3. At inclusion, patients should retrospectively have from 2 to 8 migraine attacks per month during the last 3 months. This frequency must be confirmed in the headache diary before randomization to treatment.
4. Debut of migraine at least one year prior to inclusion
5. Start of migraine before age 50 years
6. No use of other migraine prophylactics during the study
7. For women of child-bearing potential, use of highly effective contraception.

Exclusion Criteria:

1. Interval headache not distinguishable from migraine;
2. Chronic migraine, chronic tension-type headache, medication overuse headache or other headache occurring on ≥ 15 days/month
3. Pregnancy, planning to get pregnant, inability to use contraceptives, lactating
4. Clinical information on or signs of cholestasis or decreased hepatic or renal function. If in doubt, relevant blood tests should be performed
5. High degree of comorbidity and/or frailty associated with reduced life expectancy or high likelihood of hospitalization, at the discretion of the investigator
6. Hypersensitivity to candesartan
7. History of angioneurotic oedema
8. Current use of antihypertensive medication
9. Current use of potassium supplements
10. Current use of spironolactone
11. Primary hyperaldosteronism (Conn's syndrome)
12. Significant psychiatric illness
13. Use of medicines for migraine prophylaxis less than 4 weeks, or of botulinum toxin less than 16 weeks, prior to start of study
14. Having tried ≥ 3 prophylactic drugs against migraine during the last 10 years
15. Previous use of candesartan
16. Requiring detoxification from acute medication (triptans, opioids)
17. Consistently failing to respond to any acute migraine medication
18. Alcohol or illicit drug dependence.
19. Inability to understand study procedures and to comply with them for the entire length of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-08-08 (Actual)

PRIMARY OUTCOMES:
change in number of migraine days per 4 weeks, from baseline | 20 weeks plus final visit 1 week after treatment
  participants will fill in a headache diary during 20 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Samsonsen, md phd, Study Director — St Olavs Hospital, Dept Neurology & Clinical Neurophysiology; Jorunn L Helbostad, prof, Study Director — Norwegian University of Science and Technology, Fac MH, Dept INB; Erling Tronvik, md prof, Principal Investigator — Norwegian University of Science and Technology, Fac MH, Dept INB
Locations (10):
- Tartu University Clinics, Tartu, Estonia
- Norway (9):
  - Haukeland University Hospital, Bergen
  - Nordland Hospital, Bodø
  - Sørlandet Hospital, Kristiansand
  - Akershus University Hospital AHUS, Lørenskog
  - Møre and Romsdal Hospital Molde, Molde
  - Rikshospitalet University Hospital, Oslo
  - Ullevål University Hospital, Oslo
  - University Hospital of North Norway, Tromsø
  - St Olavs Hospital, Trondheim

REFERENCES:
- [Derived] Oie LR, Wergeland T, Salvesen O, Gravdahl GRB, Aschehoug I, Gulati S, Bj Rk MH, Lundqvist C, Alstadhaug KBR, Winsvold BS, Aamodt AH, Larsen IC, B E MG, Braschinsky M, Muller B, Vetvik KGT, Muller KI, Aaseth K, Khanevski AN, Ovrevik AB, Vegrim HM, Lindroos J, Eid K, Engstrand H, Bezgal B, Larsen MB, Osthus JHG, Stovner LJ, Tronvik E. Candesartan versus placebo for migraine prevention in patients with episodic migraine: a randomised, triple-blind, placebo-controlled, phase 2 trial. Lancet Neurol. 2025 Oct;24(10):817-827. doi: 10.1016/S1474-4422(25)00269-8. PMID 40975098